CLINICAL TRIAL: NCT00166920
Title: Measurement of Cerebral Oxygen Extraction Fraction Using MRI Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701261
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
All images in this study were acquired on a 1.5 T Sonata whole body scanner (Siemens Medical Inc., Erlangen, Germany) using 2D multi-echo gradient echo/spin echo sequence and 2D single-shot gradient echo-planar imaging sequence plus intravenous magnetic susceptibility contrast medium. The quantitative estimates and mapping of cerebral metabolic rate of oxygen utilization were calculated and plotted in all subjects.

DETAILED DESCRIPTION:
All images in this study were acquired on a 1.5 T Sonata whole body scanner (Siemens Medical Inc., Erlangen, Germany) using 2D multi-echo gradient echo/spin echo sequence and 2D single-shot gradient echo-planar imaging sequence plus intravenous magnetic susceptibility contrast medium. The quantitative estimates and mapping of cerebral metabolic rate of oxygen utilization were calculated and plotted in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* normal volunteer
* stroke

Exclusion Criteria:

* who is unable receiving MRI examination
* pregnancy

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2004-07; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Man Liu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Province of Taiwan, Taiwan